CLINICAL TRIAL: NCT05269901
Title: Association Between GPX4 Dependent Ferroptosis Pathway and Epilepsy in School-aged Children
Brief Title: Association Between Ferroptosis and Epilepsy
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/2/21
Record Dates: First submitted 2022-02-23; First posted 2022-03-08 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy
Keywords: school-aged children; ferroptosis; epilepsy; GPX4
MeSH Terms: conditions — Epilepsy | interventions — Phospholipid Hydroperoxide Glutathione Peroxidase; Genes, p53

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — school-aged children peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seizures group: 20 newly diagnosed untreated school-aged children from Jan 20, 2021 to Jan 1, 2022 in affiliated Hospital of Jiangnan University, department of pediatrics.
  Interventions: Genetic: SLC7A11, GPX4, P53
- Healthy control group: 20 age-matched healthy school-aged children from Jan 20, 2021 to Jan 1, 2022 in affiliated Hospital of Jiangnan University, department of pediatrics.
  Interventions: Genetic: SLC7A11, GPX4, P53

INTERVENTIONS:
Genetic: SLC7A11, GPX4, P53 — Obtained patients or healthy controls peripheral blood , used Western blot and Rt-qPCR to investigate the possible difference between two groups

SUMMARY:
Epilepsy is one of the most common neurologic disorders seen in children, often characterized by recurring seizures. Nearly 10.5 million children worldwide are estimated to have active epilepsy. Children with epilepsy are more likely to have developmental health and developmental comorbidities such as depression, anxiety, attention deficit hyperactivity disorder, learning disabilities, and developmental delay compared to children without epilepsy. Status epilepticus (SE) is the most common life-threatening emergency neurological emergency in children and leads to hippocampal neuronal cell death. The animal model proved SE-induced neuronal cell death in hippocampal CA1 and CA3 regions. Classical drugs like carbamazepine or phenytoin often cause behavioral problems and side effects such as unsteady gait, depression, and irritability. In addition, classical medicine did not protect cognitive function and preferred to drive drug-resistant. Therefore, it is necessary to develop a novel therapy to treat epilepsy. Ferroptosis is a new type of cell death, usually accompanied by a large amount of iron accumulation and lipid peroxidation. It is widely accepted that glutamate-mediated neuronal hyperexcitation plays a causative role in eliciting seizures, and cystine/glutamate antiporter inhibition induces ferroptosis. Hence, investigators hypothesize GPX4 dependent ferroptosis pathway may play a key role in eliciting seizures.

DETAILED DESCRIPTION:
To investigate the possible association between GPX4 dependent ferroptosis pathway and epilepsy. Investigators first obtained gene expression of GSE25453 from GEO (https://www.ncbi.nlm.nih.gov/geo), which contained ten medial temporal lobe epilepsy and ten adjacent non-seizure region tissues. Then, investigators further the possible association between GPX4 dependent ferroptosis pathway and epilepsy in school-aged children. Investigators obtained peripheral blood from 20 newly diagnosed untreated school-aged children (6 -12 years) and 20 age-matched healthy controls. Three glutathione peroxidase 4 (GPX4）dependent ferroptosis pathway biomarkers were investigated: Solute Carrier Family 7 Member 11（SLC7A11), GPX4, tumor protein 53 (P53). Western blot and Rt-qPCR were used to investigate the possible changes in these three biomarkers.

ELIGIBILITY:
Seizure group

Inclusion Criteria:

1. Aged between 6 and 12 years old
2. Newly diagnosed untreated epilepsy

Exclusion Criteria:

1. Treated with medicine or another therapy
2. Had history of cancer diseases
3. Had history of endocrine diseases

Healthy control group

Inclusion Criteria:

1. Aged between 6 and 12 years old

Exclusion Criteria:

1. Had history of epilepsy
2. Had history of cancer diseases
3. Had history of endocrine diseases

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school-aged children who admitted to our hospital from Jan 20, 2021 to Jan 1, 2022
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Rt-qPCR | Participants' blood samples were collected when enrolled in this study, and the results of different relative mRNA expression (GPX4, SLC7A11, P53) on two groups would be reported through study completion, an average of 1 year.
  Rt-qPCR allows the investigation of gene expression changes; investigators used primers as follow:
  GPX4 Forward: GAGGCAAGACCGAAGTAAACTAC GPX4 Reverse: CCGAACTGGTTACACGGGAA P53 Forward: AACTGCGGGACGAGACAGA P53 Reverse: AGCTTCAAGAGCGACAAGTTTT SLC7A11 Forward: TCTCCAAAGGAGGTTACCTGC SLC7A11 Reverse: AGACTCCCCTCAGTAAAGTGAC

SECONDARY OUTCOMES:
Western blot | Participants' blood samples were collected when enrolled in this study, and the results of different relative protein expressions (GPX4, SLC7A11, TP53) on two groups would be reported through study completion, an average of 1 year.
  Western blotting is an important technique used in cell and molecular biology. Using a western blot, investigators could investigate the possible protein differences of three GPX4 dependent ferroptosis pathway biomarkers: GPX4, SLC7A11, P53.

CONTACTS AND LOCATIONS:
Overall Officials: YueYing Liu, Study Director — Affiliated Hospital of JiangNan University, department of pediatrics
Locations (1):
- Affiliated Hospital of JiangNan University, Department of Pediatrics, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Ferroptosis is a new type of cell death, usually accompanied by a large amount of iron accumulation and lipid peroxidation. It is widely accepted that glutamate-mediated neuronal hyperexcitation plays a causative role in eliciting seizures, and cystine/glutamate antiporter inhibition induces ferroptosis. Hence, we hypothesis GPX4 dependent ferroptosis pathway may play a key role in eliciting seizures.